CLINICAL TRIAL: NCT01533090
Title: Evaluation of Reduced-volume PEG Bowel Preparation Administered the Same Day of Colonoscopy
Acronym: LowVolumePEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PMF 105
Record Dates: First submitted 2012-02-07; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2010-03

CONDITIONS: Colonic Polyps; Cancer Colon; Inflammatory Bowel Disease
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms; Inflammatory Bowel Diseases | interventions — Polyethylene Glycols; Bisacodyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- polyethylene glycol (PEG) (Active Comparator)
  Interventions: Drug: polyethylene glycol (PEG)
- PEG low volume with bisacodyl (Experimental)
  Interventions: Drug: PEG low volume with bisacodyl

INTERVENTIONS:
Drug: polyethylene glycol (PEG) — SELG-ESSE 1000 4 L: 2L THE DAY BEFORE OF COLONOSCOPY AND 2 L THE SAME DAY OF COLONOSCOPY
  Arms: polyethylene glycol (PEG)
Drug: PEG low volume with bisacodyl — Lovolesse + Lovoldyl 2L of Lovolesse with 2 or 3 tablets of bisacodyl the day before of colonoscopy or 2L of Lovolesse with 2 or 3 tablets of bisacodyl the same day of colonoscopy
  Arms: PEG low volume with bisacodyl

SUMMARY:
The conventional total dose of 4 L of polyethylene glycol (PEG) given the day before the procedure is safe and effective. It has been the standard cleansing regimen for the last 25 years. To overcome the difficulty in completing the bowel preparation due to large volume and/or taste, reduced-volume (mixed) bowel preparation of bisacodyl and 2 L of PEG have been shown to provide adequate colon cleansing and better tolerability.

LoVol-esse is a reduced-volume PEG-based bowel preparation to be used in combination with bisacodyl and designed to improve patient tolerability and attitude toward bowel cleansing prior to colonoscopy thanks to the reduced volume and improved taste. The present study is intended to compare the new dosing regimen of the bowel lavage solution given the same day compared with standard PEG formulation (SELG 1000) given the day before colonoscopy.

DETAILED DESCRIPTION:
A polyethylene glycol (PEG) electrolyte lavage solution (PEG-ELS) was originally developed in 1980 by the Fordtran group as isosmotic preparation for minimal water and electrolyte exchange with plasma to ensure safe cleansing of the bowel through a mechanical effect of large-volume lavage. The conventional total dose of 4 L given the day before the procedure is safe and effective and has been the standard cleansing regimen for the last 25 years. To overcome the difficulty in completing the bowel preparation due to large volume and/or taste, reduced-volume (mixed) bowel preparation of bisacodyl and 2 L of PEG-ELS have been shown to provide adequate colon cleansing and better tolerability.

In the last recent years, time of preparation has been demonstrated to be a critical factor for bowel preparation for colonoscopy. Several studies have demonstrated that reducing the time interval between the completion of bowel preparation and the exam improves colon cleansing compared with standard dose regimen of the PEG-electrolyte solution given the day before colonoscopy. At the same time manufacturers have tried to improve the taste and palatability of PEG formulations by adding suitable ingredients such as ascorbic acid or citric acid. LoVol-esse is a reduced-volume PEG-based bowel preparation to be used in combination with bisacodyl and designed to improve patient tolerability and attitude toward bowel cleansing prior to colonoscopy thanks to the reduced volume and improved taste. The present study is intended to compare the new dosing regimen of the bowel lavage solution given the same day compared with standard PEG formulation (SELG 1000) given the day before colonoscopy.

The results of this study will tells us if the last-hour preparation is effective and offers adequate tolerability and compliance to be adopted in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* aged between 18 and 85 yr
* undergoing a complete colonoscopy

Exclusion Criteria:

* known or suspected gastrointestinal obstruction or perforation
* toxic megacolon
* major colonic resection
* pregnant or at risk of becoming pregnant women
* lactating women
* inability to comprehend the full nature and purpose of the study
* no signed informed consent prior to inclusion in the study
* known or suspected hypersensitivity to the active principles or other ingredients
* history of anaphylaxis to drugs or allergic reactions in general

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the overall quality of bowel preparation | 4 months
  Quality of preparation will be graded according to the Ottawa Scale.

SECONDARY OUTCOMES:
safety | 4 months
  incidence and severity of the following GI unexpected adverse events: nausea, abdominal bloating, abdominal pain/cramps on a 5-point Likert scale
compliance | 4 months
  Proportion of patients able to:
  * drink < 75% of the solution (poor compliance)
  * drink at least 75% of the solution (good compliance)
  * drink all the solution (optimal compliance)

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Endoscopy Unit of Catholic University, Rome, Italy, Italy